CLINICAL TRIAL: NCT00049777
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Prophylactic Heparin in Patients With Severe Sepsis and Higher Disease Severity Who Are Undergoing Treatment With Drotrecogin Alfa (Activated)
Brief Title: A Trial of Heparin in Patients With Severe Sepsis Who Are Undergoing Treatment With Drotrecogin Alfa (Activated)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6743; F1K-MC-EVBR
Record Dates: First submitted 2002-11-13; First posted 2002-11-15 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — drotrecogin alfa activated; Heparin; Heparin, Low-Molecular-Weight

INTERVENTIONS:
Drug: Drotrecogin Alfa (Activated)
Drug: Unfractionated heparin
Drug: Low molecular weight heparin

SUMMARY:
The purpose of this study is to evaluate the relative efficacy and safety of prophylactic heparin co-administration during drotrecogin alfa (activated) infusion in the treatment of severe sepsis in the adult.

ELIGIBILITY:
Inclusion Criteria

* Adults greater than or equal to 18 years of age
* Receiving inpatient treatment for severe sepsis
* Indicated for treatment with Drotrecogin Alfa (Activated) under approved label in the country where the patient is enrolled

Exclusion Criteria

* Contraindicated for heparin treatment
* Require a higher dose of heparin than defined in the trial
* Have acute or chronic renal failure with an estimated creatinine clearance less than 30mL/min
* Weigh more than 135 kg (297 pounds)
* Are not expected to survive 28 days given their medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2002-12; Study Completion 2005-08

PRIMARY OUTCOMES:
Demonstrate in adult patients with severe sepsis who are receiving drotrecogin alfa (activated) that concomitant treatment with heparin is equivalent to treatment with placebo as determined by 28-day all-cause mortality.

SECONDARY OUTCOMES:
Determine the incidence of venous thrombotic events in patients receiving heparin vs. placebo through study days 6
and 28. Evaluate the safety profile of drotrecogin alfa (activated) and prophylactic heparin co administration by the incidence of intracranial hemorrhage and other serious bleeding events through study day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician, Berlin, Germany

REFERENCES:
- [Derived] Levi M, Levy M, Williams MD, Douglas I, Artigas A, Antonelli M, Wyncoll D, Janes J, Booth FV, Wang D, Sundin DP, Macias WL; Xigris and Prophylactic HepaRin Evaluation in Severe Sepsis (XPRESS) Study Group. Prophylactic heparin in patients with severe sepsis treated with drotrecogin alfa (activated). Am J Respir Crit Care Med. 2007 Sep 1;176(5):483-90. doi: 10.1164/rccm.200612-1803OC. Epub 2007 Jun 7. PMID 17556722